CLINICAL TRIAL: NCT06032377
Title: Improving Sleep to Protect Brain Health in Older Adults: Assessing a Novel Cognitive-behavioral Program for Insomnia Using a Multidomain Web Platform
Brief Title: Online COgnitive Behavioural Therapy for Sleep and Mental Health for Older Adults With Insomnia and Subjective Cognitive Complaints
Acronym: e-COSMOS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre de Recherche de l'Institut Universitaire de Geriatrie de Montreal (Other)
Responsible Party: Principal Investigator, Thien Thanh Dang-Vu, Professor, Neurologist; Director, Sleep, Cognition & Neuroimaging Laboratory (SCNLab), Centre de Recherche de l'Institut Universitaire de Geriatrie de Montreal
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BH210177
Record Dates: First submitted 2023-08-24; First posted 2023-09-13 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Insomnia
Keywords: insomnia; cognition; mental health; subjective cognitive complaint; sleep; online CBT; older adults; anxiety; depression; executive functions; electroencephalography; magnetic resonance imaging
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Psychological Well-Being; Anxiety Disorders; Depression | interventions — Cognitive Behavioral Therapy; Sleep

STUDY DESIGN:
Intervention Model Description: Participants with insomnia and subjective cognitive complaint are randomized into 2 groups with a 1:1 allocation ratio, after the pre-treatment assessment. Allocation will be stratified based on a composite mental health score and hypnotic medication intake. Follow-up assessments will occur 10 weeks and 24 weeks after the start of the intervention.
  One group will receive the online CBT for sleep and mental health after the baseline assessment and the other group will receive the control intervention. The group receiving the control intervention will access the CBT intervention after completion of the study.
  A good sleepers group, matched on age and gender, will also be recruited and assessed at baseline only to provide a normative reference group.
  A subgroup of participants from the insomnia group and the good sleepers group will undergo MRI and classical neuropsychological testing at baseline and 24 weeks after the start of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- online cognitive behavioral therapy for insomnia, anxiety and depression (Experimental): 10 self-directed modules of cognitive behavioral therapy for insomnia, anxiety and depression, delivered online, once a week
  Interventions: Behavioral: cognitive behavioral therapy for sleep, anxiety, and depression
- online intervention on nutrition and communication in older age (Active Comparator): 10 self-directed modules on healthy nutrition habits and communication strategies, delivered online, once a week
  Interventions: Behavioral: education about healthy nutrition habits and communication in older age

INTERVENTIONS:
Behavioral: cognitive behavioral therapy for sleep, anxiety, and depression — This intervention addresses insomnia, anxiety and depression via modules covering all the core CBTi components: psychoeducation about insomnia, relaxation, cognitive restructuring, stimulus control, sleep restriction and stress management; as well as psychoeducation about anxiety and low mood, behavioral activation strategies, and strategies to better manage ruminations. The modules are adapted to older adults and include short texts, pictures, quizzes with feedback, interactive exercises, logbooks, audio and video recordings.
  Other Names: eCBTi+
  Arms: online cognitive behavioral therapy for insomnia, anxiety and depression
Behavioral: education about healthy nutrition habits and communication in older age — This intervention addresses healthy nutrition habits as well as communication and aging. The modules are adapted to older adults and include short texts, pictures, quizzes with feedback, interactive exercises, logbooks, audio and video recordings
  Other Names: active control
  Arms: online intervention on nutrition and communication in older age

SUMMARY:
The goal of this randomized controlled clinical trial is to assess a novel cognitive-behavioral program for sleep and mental health using a multidomain web platform (eCBTi+) in participants with insomnia and subjective cognitive complaint. The main questions it aims to answer are:

* Whether the eCBTi+ intervention improves sleep (subjective: Insomnia severity index [ISI], objective: EEG-based sleep efficiency) sleep and mental health (Geriatric Anxiety Index [GAI] and Geriatric Depression Scale [GDS]) compared to the control intervention
* Whether the eCBTi+ intervention improves cognitive abilities (subjective: Cognitive Failure Questionnaire [CFQ], objective: CANTAB executive functions composite score) compared to the control intervention

DETAILED DESCRIPTION:
Participants with insomnia disorder will complete:

* A phone interview
* Two video conferences (assessment of eligibility and tutorial to set up sleep monitoring devices)
* 9 nights of at-home polysomnography with an EEG headband (3 times x 3 nights)
* 42 sleep diaries (3 times x 14 days)
* 42 days wearing an actigraphy device (3 times x 14 days)
* Online questionnaires
* Phone call for a check-in with a psychologist
* 3 cognitive testing sessions
* 10 modules of online information on health, over the course of 10 weeks
* In MRI subgroup: 2 in-person testing

Good sleeper participants will complete:

* A phone interview
* Two video conferences (assessment of eligibility and tutorial to set up sleep monitoring devices)
* 3 nights of at-home polysomnography with an EEG headband
* 14 sleep diaries
* 14 days wearing an actigraphy device
* Online questionnaires
* 1 cognitive testing session
* 1 in person session for MRI.

In addition, researchers will compare outcomes from participants with insomnia and subjective cognitive complaint to a group of good sleepers to have normative values for imaging data.

ELIGIBILITY:
Inclusion

* age 60 years or older at the time of enrolment
* Sleep Condition Indicator, SCI ≤ 16 and/or meeting DSM-V criteria based on the symptoms assessed by the SCI
* subjective cognitive complaints (self-report version of Everyday Cognition scale (ECog), score ≥ 2 on any item)
* ability to read and understand French or English
* ability to use a smartphone or tablet, and access to home internet connection
* If on hypnotic or psychotropic medication (including cannabis), being on stable dosage for at least 2 months prior to study entry
* Score on the STOP-BANG questionnaire < 3 corresponding to participants with low risk of obstructive sleep apnea

Exclusion

* located outside of Québec or Ontario
* current hospitalization or planned major surgery
* uncorrected severe hearing or vision impairment
* reported diagnosis of major neurocognitive disorder or mild cognitive impairment (MCI)
* performance suggestive of major neurocognitive disorder or MCI on T-MoCA < 17
* reported diagnosis of schizophrenia or bipolar disorder
* reported diagnosis or positive screen on the MINI for psychotic or bipolar disorders
* high suicidal risk, as assessed by the modified Columbia-Suicide Severity Rating Scale
* reported diagnosis or positive screening (apnea-hypopnea index >30 on a level 3 home sleep apnea test) for another untreated sleep disorder (e.g., sleep disordered breathing (OSA), REM sleep behavior disorder (RBD), restless legs syndrome (RLS); individuals with treated and controlled OSA (residual apnea-hypopnea index <30 and good therapeutic compliance) or RLS will not be excluded
* current shift work
* currently receiving CBT, having received CBTi in the past
* frequent alcohol consumption having an impact on functionning (>10 glasses/week and having a significant impact on functionning)
* illicit drugs use (more than once a month)

Additional exclusion criteria for neuroimaging

* psychotropic (including hypnotic) medication in the past 2 weeks
* contraindications for MRI (e.g., pacemaker, metallic implant, claustrophobia)
* unable or unwilling to come to one of the participating MRI centers (Montreal, Ottawa)
* medical conditions likely to affect sleep; in particular:
* current neurological disorder (e.g., epilepsy with any seizure in the past year, concussion in the past 3 months, multiple sclerosis, Parkinson's disease)
* past history of brain lesion (e.g., brain hemorrhage, brain tumor, any condition having required brain surgery)
* major surgery (i.e., requiring general anesthesia) in the past 3 months
* untreated thyroid disorder
* chronic pain syndrome self-reported as interfering with sleep (e.g., migraine, fibromyalgia, rheumatoid arthritis)
* recent and severe infection in the past 3 months (e.g., pneumonia, kidney infection)
* active cancer or treated cancer with post-cancer treatment for less than 2 years

Inclusion/exclusion criteria for good sleepers Twenty-five good sleepers without cognitive complaint will be recruited as controls for the MRI session following the same criteria described above, except that SCI ≥ 17, not meeting the diagnostic criteria for chronic insomnia as assessed by the insomnia module of the SCID and no subjective cognitive complaint.

Ages: 60 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 275 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Insomnia severity index | At baseline, at 10-12 weeks and at 24 weeks after the start of the intervention
  Change in Insomnia Severity Index. ISI range from 0 to 28, higher score means more severe insomnia symptoms.
Subjective cognitive impairment based on cognitive failure questionnaire | At baseline, at 10-12 weeks and at 24 weeks after the start of the intervention
  Change in Cognitive Failure Questionnaire (CFQ) total score as well as number of items with a score ≥ 3. The CFQ comprises 25 items and total score corresponds to the sum of all completed items, total score range from 0 to 100.
Objective cognitive performance based on a composite score for executive functions from the CANTAB | At baseline and at 24 weeks after the start of the intervention
  Change in the Cambridge Neuropsychological Test Automated Battery (CANTAB) executive functions composite score (Intra-Extra Dimensional Set Shift [IED] and Stocking of Cambridge [SOC], ranging from 0 to 100 with higher scores reflecting poorer executive functions.
Geriatric anxiety index | At baseline, at 10-12 weeks and at 24 weeks after the start of the intervention
  Change in Geriatric anxiety index. GAI scores range from 0 to 20 and higher scores mean more severe anxiety symptoms.
Geriatric depression scale | At baseline, at 10-12 weeks and at 24 weeks after the start of the intervention
  Change in Geriatric depression scale. GDS scores range from 0 to 15, higher scores mean more severe depression symptoms.

SECONDARY OUTCOMES:
Sleep quality based on the Pittsburgh sleep quality index | At baseline, at 10-12 weeks and at 24 weeks after the start of the intervention
  Change in Pittsburgh sleep quality index. PSQI scores range from 0 to 21, higher scores mean worse sleep quality.
Objective sleep measures based on actigraphy: Sleep Efficiency | At baseline, at 10-12 weeks and at 24 weeks after the start of the intervention
  Change in Sleep Efficiency (SE) from actigraphs. Sleep efficiency ranges from 0 to 100, values closer to 100 mean greater sleep efficiency.
Objective sleep measures based on actigraphy: Sleep Latency | At baseline, at 10-12 weeks and at 24 weeks after the start of the intervention
  Change in Sleep Latency (SL) from actigraphs. Sleep latency in minutes, greater values mean longer time to fall asleep.
Objective sleep measures based on actigraphy: Total Sleep Time | At baseline, at 10-12 weeks and at 24 weeks after the start of the intervention
  Change in Total Sleep Time (TST) from actigraphs. Total Sleep Time in minutes, greater values mean longer time spent asleep.
Objective sleep measures based on actigraphy: Wake After Sleep Onset | At baseline, at 10-12 weeks and at 24 weeks after the start of the intervention
  Change in Wake After Sleep Onset (WASO) from actigraphs. Wake After Sleep Onset in minutes, greater values mean longer time spent awake.
Objective sleep measures based on EEG: Sleep Efficiency | At baseline, at 10-12 weeks and at 24 weeks after the start of the intervention
  Change in Sleep Efficiency (SE) from EEG. Sleep efficiency ranges from 0 to 100, values closer to 100 mean greater sleep efficiency.
Objective sleep measures based on EEG: Sleep Latency | At baseline, at 10-12 weeks and at 24 weeks after the start of the intervention
  Change in Sleep Latency (SL) from EEG. Sleep latency in minutes, greater values mean longer time to fall asleep
Objective sleep measures based on EEG: Total Sleep Time | At baseline, at 10-12 weeks and at 24 weeks after the start of the intervention
  Change in Total Sleep Time (TST) from EEG. Total Sleep Time in minutes, greater values mean longer time spent asleep.
Objective sleep measures based on EEG: Wake After Sleep Onset | At baseline, at 10-12 weeks and at 24 weeks after the start of the intervention
  Change in Wake After Sleep Onset (WASO) from EEG. Wake After Sleep Onset in minutes, greater values mean longer time spent awake.
Objective sleep measures based on EEG: Slow Wave Activity | At baseline, at 10-12 weeks and at 24 weeks after the start of the intervention
  Change in Slow Wave Activity (SWA) power density from EEG.
Objective sleep measures based on EEG: Slow Wave Sleep | At baseline, at 10-12 weeks and at 24 weeks after the start of the intervention
  Change in Slow Wave Sleep (SWS) from EEG. Slow Wave Sleep in minutes, greater values mean longer time spent in Slow Wave Sleep.
Subjective sleep measures based on sleep diaries: Sleep Efficiency | At baseline, at 10-12 weeks and at 24 weeks after the start of the intervention
  Change in Sleep Efficiency (SE) from sleep diaries. Sleep efficiency ranges from 0 to 100, values closer to 100 mean greater sleep efficiency.
Subjective sleep measures based on sleep diaries: Sleep Latency | At baseline, at 10-12 weeks and at 24 weeks after the start of the intervention
  Change in Sleep Latency (SL) from sleep diaries. Sleep latency in minutes, greater values mean longer time to fall asleep.
Subjective sleep measures based on sleep diaries: Total Sleep Time | At baseline, at 10-12 weeks and at 24 weeks after the start of the intervention
  Change in Total Sleep Time (TST) from sleep diaries. Total Sleep Time in minutes, greater values mean longer time spent asleep.
Subjective sleep measures based on sleep diaries: Wake After Sleep Onset | At baseline, at 10-12 weeks and at 24 weeks after the start of the intervention
  Change in Wake After Sleep Onset (WASO) from sleep diaries. Wake After Sleep Onset in minutes, greater values mean longer time spent awake.
Cognitive performances from the CANTAB: Rapid Visual Information Processing (RVP) | At baseline, at 10-12 weeks and at 24 weeks after the start of the intervention
  Change in Rapid Visual Information Processing RVP - A' (sensitivity to the target sequence) and probability of false alarm (range: 0.00 - 1.00; bad to good)].
Cognitive performances from the CANTAB: Spatial Span (SSP) | At baseline, at 10-12 weeks and at 24 weeks after the start of the intervention
  Change in Spatial Span [SSP - Forward/Reverse Span Lengths (range: 2-9; bad to good]
Cognitive performances from the CANTAB: Spatial Working Memory (SWM) | At baseline, at 10-12 weeks and at 24 weeks after the start of the intervention
  Change in Spatial Working Memory [SWM - Number of times the subject incorrectly revisits a box in which a token has previously been found (range: 0 - ∞; good to bad)].
Cognitive performances from the CANTAB: Paired Associates Learning (PAL) | At baseline, at 10-12 weeks and at 24 weeks after the start of the intervention
  Change in Paired Associates Learning [PAL - Total errors adjusted (range: 0 - 70; good to bad; First attempt memory score (range: 0-20; bad to good)]
Cognitive performances from the CANTAB: Pattern Recognition Memory (PRM) | At baseline, at 10-12 weeks and at 24 weeks after the start of the intervention
  Change in Pattern Recognition Memory [PRM - Percent correct immediate/delayed (range: 0-100; bad to good)].
Cognitive performances from the CANTAB: Intra-Extra Dimensional Set Shift (IED) | At baseline, at 10-12 weeks and at 24 weeks after the start of the intervention
  Intra-Extra Dimensional Set Shift, IED - number of times that the subject failed to select the stimulus compatible with the current rule on the stage where the extra-dimensional shift occurs (range: 0-50; good to bad); Total errors adjusted (range: 0-402; good to bad)
Cognitive performances from the CANTAB: Stocking of Cambridge (SOC) | At baseline, at 10-12 weeks and at 24 weeks after the start of the intervention
  Stocking of Cambridge, SOC - Number of problems successfully completed in the minimum possible number of moves (range: 0 - 12; bad to good); Mean number of moves required to complete problems (range: 5 - 12; good to bad); Initial thinking time median (range: 0 ms to ∞; longer times may indicate better planning efforts
Negative emotional bias measured on the Cambridge Neuropsychological Test Automated Battery (CANTAB) | At baseline, at 10-12 weeks and at 24 weeks after the start of the intervention
  Change in Emotional Bias Task (EBT) subscales from the CANTAB [EBT - proportion of trials rated as 'Happy' (range: 0-15, bad to good)].
Memory encoding fMRI activations | At baseline, at 24 weeks after the start of the intervention
  Change in fMRI activation level (arbitrary units) in the hippocampus, temporal lobe and prefrontal cortex during the memory encoding task.
Cognitive performance (classical neuropsychological tests) | At baseline, at 24 weeks after the start of the intervention
  all subscales from classical neuropsychological test battery (Trail Making Test A [TMT-A], Digit Symbol Substitution test (WAIS), Boston Naming Test, Digit Span - forward and backward (WAIS), Rey Auditory Verbal Learning test, Logical Memory I and II (Wechsler Memory Scale), Brief Visuospatial Memory Test Revised (BVMT-R), Trail Making Test B [TMT-B], Verbal Fluency Test (from D-KEFS), Color-Word Interference Test [Stroop test, from D-KEFS]).
Cortical thickness measures | At baseline, at 24 weeks after the start of the intervention
  Change in cortical thickness (mm) in the prefrontal cortex and precuneus.
Fractional anisotropy | At baseline, at 24 weeks after the start of the intervention
  Change in fractional anisotropy of the superior longitudinal fasciculus and internal capsule.
Resting-state measures | At baseline, at 24 weeks after the start of the intervention
  Change in the ratio between segregation and integration within and between the default-mode network and the limbic network during resting-state as measured with functional connectivity.
GABA/glutamate ratio from magnetic resonance spectroscopy | At baseline, at 24 weeks after the start of the intervention
  Change in the GABA/glutamate ratio in the anterior cingulate cortex.
Treatment-mediated association between changes in sleep and cognition | At 10-12 weeks and at 24 weeks after the start of the intervention
  Mediation estimate of the extent to which exposure to eCBTi+ explains the association between improved sleep and improved cognition
Satisfaction from System Usability Scale | At 10-12 weeks after the start of the intervention
  Score on the System Usability Scale, reflecting the degree to which participants were satisfied with the eCBTi+ and the control intervention. Percentage ranging between 0 and 100%.
Technology acceptance | At 10-12 weeks after the start of the intervention
  Score on the extended version of the Technology Acceptance Model-2 reflecting th degree to which participants use and intend to use the eCBTi+ (and control intervention) as implemented on e-SPACE. Each process influencing technology acceptance is scored on a 7-point Likert scale.
Adherence to treatment | At 10-12 weeks after the start of the intervention
  Number of modules completed as a measure of treatment adherence

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - The Royal's Institute of Mental Health Research (IMHR), Ottawa, Ontario
  - Centre intégré universitaire de santé et de services sociaux du Centre-Sud-de l'Île-de-Montréal. CCSMTL - IUGM, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Undecided